CLINICAL TRIAL: NCT00291005
Title: A Multicenter Phase II Open Label Non-Comparative Trial of RP56976 Administered Every Three Weeks in Combination With Daily Prednisolone for Metastatic Hormone Refractory Prostate Cancer
Brief Title: PhII One Label Non-Comparative Trial in Metastatic Hormone Refractory Prostate Cancer in Combination With Prednisolone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARD6562; XRP6976J/2101
Record Dates: First submitted 2006-02-10; First posted 2006-02-13 (Estimated); Last update posted 2009-03-27 (Estimated); Status verified 2009-03

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate cancer; HRPC; AIPC; Hormone refractory; Androgen independent; Docetaxel; Taxotere; prednisolone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel

INTERVENTIONS:
Drug: ARD6562, Docetaxel

SUMMARY:
* To evaluate the overall tumor response rate in subjects with metastatic hormone refractory prostate cancer
* To evaluate PSA (tumor marker) response rate
* To evaluate safety

ELIGIBILITY:
Inclusion Criteria:

* Men with prostate adenocarcinoma with at least one metastatic lesion which is measurable and who progressed after prior hormonal therapy.

Exclusion Criteria:

* 1.Body temperature > 38 degree centigrade.
* 2.Prior radiotherapy to > 25% of bone marrow.
* 3.Prior isotope therapy and/or brachytherapy
* 4.Prior gene therapy.
* 5.Active double cancer.
* 6.Known brain or leptomeningeal involvement.
* 7.History of hypersensitivity reaction to drug
* 8.Other serious illness or medical condition
* 9.Subjects whom the investigators consider inappropriate from social or medical aspects.

Ages: 20 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42
Dates: Start 2004-08

PRIMARY OUTCOMES:
Overall tumor response rate by Response Evaluation Criteria in Solid Tumor (RECIST)

SECONDARY OUTCOMES:
Overall response rate by modified WHO criteria, PSA response rate, safety

CONTACTS AND LOCATIONS:
Overall Officials: Atsushi NAKAMURA, Study Chair — CSD, PL / TA-Oncology
Locations (1):
- Sanofi-Aventis, Tokyo, Japan